CLINICAL TRIAL: NCT04520815
Title: Assessment of the Prevalence and Kinetics of Diaphragmatic Dysfunction in Elderly Patients With Acute Respiratory Distress
Brief Title: Prevalence and Kinetics of Diaphragmatic Dysfunction in Elderly Patients With Acute Respiratory Distress
Acronym: OLDIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/CHU/10
Record Dates: First submitted 2020-06-24; First posted 2020-08-20 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Respiratory Distress Syndrome, Adult
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute respiratory distress (ARD) is one of the most frequent reasons for consultation and hospitalization in emergency medicine. The use of ultrasound methods as a diagnostic and clinical assessment tool in emergency medicine is increasingly important. As such, ultrasound is a simple, non-invasive means of assessing diaphragmatic function in the patient's bed. Several methods of ultrasound assessment of diaphragm function have been described. Among these different methods, the diaphragmatic excursion seems to have a better intra and interobserver reproducibility as well as a greater feasibility, in particular because of its speed of realization and its learning curve seeming faster in comparison with the measurement. of the thickening fraction. Measuring the diaphragmatic excursion could therefore ultimately represent a simple means of assessing respiratory function, both diagnostic and prognostic, in patients with acute respiratory distress in the emergency departments. The etiologies of acute respiratory distress in very elderly patients (i.e.> 75 years) admitted to the emergency reception service are multiple.

To our knowledge, there is no data available in the literature on the prevalence of diaphragmatic dysfunction and its short- and long-term course in this category of patients. The main objective of this study is therefore to assess the prevalence of diaphragmatic dysfunction and its evolutionary kinetics in patients over the age of 75 admitted for acute respiratory distress in the emergency medicine department.

ELIGIBILITY:
Inclusion Criteria:

* Patient in spontaneous ventilation at the admission on emergency room
* Presence of acute respiratory distress defined by at least 1 of the following criteria:

  * Respiratory rate > 25/min and/or clinical signs of acute respiratory distress,
  * Hypoxia defined by Sp02 < 90 %,
  * Hypercapnia defined by PaC02 > 45 mmHg with respiratory acidosis defined by a pH value <7.35.
* Absence of opposition of the patient to his participation in the study and the use of his data or the trusted person if the state of the patient does not allow it.

Exclusion Criteria:

* Presence of a preexisting diaphragmatic dysfunction appearing in the history or the medical file of the patient and explored on the electro-physiological level,
* Patient with acute respiratory distress on arrival at the SAU with clinical criteria justifying immediate use of invasive mechanical ventilation and not allowing ultrasound measurements to be carried out or patient admitted to the SAU with mechanical ventilatory support from the outset,
* Poor command of the French language or state incompatible with the patient's understanding and / or informed adherence to the study protocol,
* History of surgery involving the integrity of the diaphragmatic muscle (diaphragm plication or diaphragmatic lumpectomy or placement of diaphragmatic pacemaker),
* Criteria for shock or severe hemodynamic instability,
* Intra-cranial hypertension.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Recruitment of all patients over the age of 75, presenting to adult emergency departments and in spontaneous ventilation and having at least one criterion of acute respiratory distress.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-24 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Presence of diaphragmatic dysfunction | inclusion
  Ultrasound measurement of diaphragmatic excursion (ED)
Presence of diaphragmatic dysfunction | Day 1
  Ultrasound measurement of diaphragmatic excursion (ED)
Presence of diaphragmatic dysfunction | Day 3
  Ultrasound measurement of diaphragmatic excursion (ED)
Presence of diaphragmatic dysfunction | Day 7
  Ultrasound measurement of diaphragmatic excursion (ED)
Presence of diaphragmatic dysfunction | up to 7 days
  Ultrasound measurement of diaphragmatic excursion (ED)

SECONDARY OUTCOMES:
Inter-observer reproductibility of the measurement of ED and EIT | Day 0
  Comparison of the measure in the between two operators
Predictive value of the presence of diaphragmatic dysfunction | 48 hours after the beginning of hospitalization
  Ultrasound measurement of diaphragmatic excursion (ED) on the use of ventilatory assistance
Predictive value of the presence of diaphragmatic dysfunction over the average length of hospital stay | up to 7 days
  length of hospitalization duration in Intensive care unit
Predictive value of the presence of a diaphragmatic dysfunction on mortality | up to 7 days
  Ultrasound measurement of diaphragmatic excursion (ED)
Predictive value of the presence of a diaphragmatic dysfunction on mortality | 6 months after the end of hospitalization
  Ultrasound measurement of diaphragmatic excursion (ED)
Kinetics of evolution of the diaphragmatic function | Day 1
  Ultrasound measurement of diaphragmatic excursion (ED)
Kinetics of evolution of the diaphragmatic function | Day 3
  Ultrasound measurement of diaphragmatic excursion (ED)
Evolution of the diaphragmatic function | Day 7
  Ultrasound measurement of diaphragmatic excursion (ED)
Evolution of the diaphragmatic function | Before 7 days
  Ultrasound measurement of diaphragmatic excursion (ED)
Correlation between risk factors for developing diaphragmatic dysfunction (DD) and ultrasound diagnosis of diaphragmatic dysfunction (DD) | up to 7 days
  Identification of the risk factors and Ultrasound measurement of diaphragmatic excursion (ED)
Possible correlation between the presence of a DD diagnosed by the ultrasound measurement of the ED and the duration of mechanical ventilation, the duration of hospitalization in ICU, respiratory complications rate and failures organs rate | up to 7 days
  qSOFA et APACHE II score
Correlation between the presence of DD diagnosed by ultrasound measurement of ED and the evolution of the functional status of the patient at the end of hospitalization compared to his status at the admission | up to 7 days
  scores ADL et AGGIR
Presence of diaphragmatic dysfunction in patients with COVID-19 | up to 7 days
  Ultrasound measurement of diaphragmatic excursion (ED)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas GROSEIL, Dr, Principal Investigator — CHU de La Réunion
Locations (1):
- Centre Hospitalier Universitaire de la Réunion, Saint-Denis, France

IPD SHARING:
Plan to Share IPD: No